CLINICAL TRIAL: NCT05932875
Title: Peanut Consumption to Augment Adaptations to Concurrent Resistance and Aerobic Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwestern University (Other)
Responsible Party: Principal Investigator, Edward Merritt, Associate Professor of Kinesiology, Southwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SP23_20
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Muscle Strength; Cardiorespiratory Fitness; Body Composition; Peanut Consumption
Keywords: peanut; muscle health; concurrent training; cardiorespiratory fitness
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut/Carbohydrate Consumption Exercise Training (Active Comparator): Participants in this group will undergo 16 weeks of concurrent exercise training (4 sessions/week) consuming a peanut-based rice/oatmilk smoothie after each workout
  Interventions: Other: Exercise Training
- Carbohydrate Consumption Exercise Training (Placebo Comparator): Participants in this group will undergo 16 weeks of concurrent exercise training (4 sessions/week) consuming a rice/oatmilk smoothie after each workout
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Exercise Training — 4 day per week concurrent exercise training program

SUMMARY:
The primary objective of this proposal is to determine the effects of post-exercise peanut consumption on long-term aerobic and resistance exercise training adaptations in middle-aged men and women. The investigators will determine the impact of peanuts on exercise training-induced improvements in muscle strength, gains in muscle mass, and improvements in cardiorespiratory fitness and metabolic capacity.

DETAILED DESCRIPTION:
Positive health benefits of peanut consumption are well-known, but potential benefits have yet to be discovered, especially in regard to fitness. This project will directly determine the benefits of peanut consumption as part of a long-term aerobic and resistance exercise training program in middle-aged adults.

Proper nutrition is necessary for the body to properly recover and adapt to an exercise bout and thereby realize the health benefits of the exercise. The period of time immediately after exercise is even more important in realizing these adaptations. With relatively higher amounts of fats, peanuts are often overlooked as a nutritious, post-exercise snack, because they might not be optimal for athletic performance. However, for a middle-aged adult performing the recommended amount of weekly physical activity, the protein and carbohydrate content of peanuts is sufficient to provide the macronutrients necessary to achieve the beneficial health adaptations associated with exercise training. Other micronutrients and healthy fats in peanuts, might confer further benefits beyond those of other post-exercise supplements, however, this has yet to be elucidated.

The randomized, placebo-controlled, clinical trial will provide valuable information on the health benefits of peanut consumption and determine if peanuts can augment beneficial exercise training adaptations in middle-aged adults. The investigators will recruit a group of 48 adults (30-55 years) who do not regularly exercise to undertake a 4-month exercise training program. The program, proven to increase muscle mass and improve cardiorespiratory fitness, will consist of 4 days per week of structured workouts (2/week resistance, 2/week aerobic). Participants will be randomly assigned to consume either a peanut-based snack or an isocaloric, non-peanut carbohydrate-based snack immediately after each exercise session. A comprehensive health and fitness assessment will be conducted before training, after 2-months of training, and after 4-months of training. Measures of cardiorespiratory fitness, muscular fitness, and body composition will be assessed.

Anticipated Products & Potential Outcomes When completed, this study will provide the first evidence of the effect of post-exercise peanut consumption on long-term exercise training adaptations to both aerobic and resistance training in middle-aged adults. This will be the first study to determine the effects of peanut consumption with aerobic exercise training, and the longest study on resistance exercise training and peanut consumption. With the mid-training 2-month timepoint, the investigators will be able to compare our results to those of similar resistance training peanut studies, but importantly follow them for longer, when resistance training adaptations are likely to be more apparent. The investigators hypothesize that the peanut group will experience greater gains in muscle strength and hypertrophy than the placebo group. The investigatorshypothesize that the peanut and placebo group will have similar improvements in cardiorespiratory fitness and body composition (higher total body lean mass leading to relatively lower body fat). This would be an important finding to prove that, despite their higher fat content, peanut consumption does not lead to negative effects on body composition nor prevent cardiorespiratory adaptions due to exercise training. Overall, the results are likely to demonstrate that peanuts are a simple, inexpensive, and effective post-exercise health food capable of further enhancing the beneficial effects of exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 30- 55 years old
* healthy
* non-smoking
* no exercise training in the previous 6 months
* not currently attempting to gain or lose weight
* body mass index < 35
* no need for physician clearance prior to beginning an exercise program as determined by American College of Sports Medicine guidelines.

Exclusion Criteria:

* neurological or musculoskeletal disorders
* uncontrolled hypertension (resting systolic blood pressure > 180 mmHg or diastolic > 120 mmHg
* unstable or exercise-induced angina pectoris
* diabetes mellitus; any other medical condition that would interfere with testing or training
* androgen (e.g., testosterone), anabolic (e.g., GH, IGF-I), or catabolic (e.g. GLP-1 agonists) therapy
* food allergy to peanuts or dairy products
* pregnant people or people actively trying to get pregnant
* on a special diet that restricts protein/carbs/sugar/fat.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Total Lean Mass | From baseline to the end of the training program at 16 weeks.
  Amount of lean mass as determined by dual energy x-ray absorptiometry scan
Muscle strength | From baseline to the end of the training program at 16 weeks.
  Isometric grip and knee extension strength, as well as dynamic 1-repitition maximum strength of bench press, leg press, overhead press, knee extension
Cardiorespiratory fitness | From baseline to the end of the training program at 16 weeks.
  Maximal oxygen consumption as determined by graded treadmill test

CONTACTS AND LOCATIONS:
Locations (1):
- Southwestern University, Georgetown, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IRB approval does not allow for IPD to be shared.